CLINICAL TRIAL: NCT03020186
Title: Effects of Green-MED Diet Via the Gut-fat-brain Axis; DIRECT-PLUS
Brief Title: Effects of Green-MED Diet Via the Gut-fat-brain Axis
Acronym: DIRECT-PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); University of Leipzig (Other)
Responsible Party: Principal Investigator, Iris Shai, Principle investigator, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BGU
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2017-01

CONDITIONS: Abdominal Obesity Metabolic Syndrome
MeSH Terms: conditions — Abdominal obesity metabolic syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Physical activity (Placebo Comparator): Physical activity (PA) group will receive free gym memberships and the instruction necessary to engage in moderate-intensity physical activity, ~80% of which will have an aerobic component. The participants will get basic health promoting guideline for healthy diet .
  Interventions: Other: Physical activity
- Physical activity+ MED diet (Experimental): On top of the PA intervention described in Arm 1, the participants will be guided for moderate weight loss with a traditional Mediterranean (MED) diet, low in simple carbohydrates. The diet will include 1oz/day of walnuts that will be provided free of charge.
  Interventions: Other: Physical activity+ MED diet
- Physical activity+ green-MED diet (Experimental): On top of the PA intervention described in Arm 1, the participants will guided for moderate weight loss with a MED diet, low in simple carbohydrates that will be rich in plants and polyphenols and low in processed meat. The diet will include 1oz/day of walnuts, 3-4 cups/day of green tea and ~500cc green shake/dinner based on specific strain of duckweed [Wolffia globose, "Mankai"], an aquatic plant, which might serve as a plant protein source. All the above will be provided free of charge.
  Interventions: Other: Physical activity+green MED diet

INTERVENTIONS:
Other: Physical activity
  Arms: Physical activity
Other: Physical activity+ MED diet
  Arms: Physical activity+ MED diet
Other: Physical activity+green MED diet — ****Sub-study from all 3 main arms: Autologous fecal microbiota supplement intervention derived from the time of maximal weight loss: At the 6-month time period, the time of anticipated greatest weight reduction, participants's feces samples will be processed to capsulized inocula. Samples will be frozen within 2 hours and will be kept at -80c pending analysis. Participants will be randomized to receive either research capsules or identical placebo capsules between 8 and 14 months time period. Placebo capsules will consist of a combination of powdered cocoa and vegetable gelatin in normal saline/glycerol and will be identical in appearance to research capsules.
  Arms: Physical activity+ green-MED diet

SUMMARY:
Mediterranean (MED) diet, richer in plants/seeds (and dietary polyphenols) and low in processed meat (green-MED diet) may have a pronounced beneficial effect on age-related declines that begin in middle age, reflected by changes in adiposity, cognitive function, and cardiometabolic risk. The investigators hypothesize that long-term intake of this diet will significantly potentiate the effects of a healthy lifestyle (physical activity and Mediterranean diet), constituting a powerful strategy to halt or even reverse the progression of several age-related processes related to adiposity, cardiometabolic health and cognition. The investigators further hypothesize that lifestyle intervention might modify the gut microbiota profile and that autologous fecal microbiota supplement derived from the time of maximal weight loss might halt the expected subsequent regain phase.

DETAILED DESCRIPTION:
The investigators aim to compare the effect of green-MED diet+ physical activity (PA) vs. MED diet+ PA vs. PA on the gut-fat-brain axis and to explore the additional contribution of autologous fecal microbiota derived at the rapid weight loss phase on regain phase. Mediterranean (MED) diet, richer in plants/seeds (and dietary polyphenols) and low in processed meat may have a pronounced beneficial effect on age-related declines that begin in middle age, reflected by changes in adiposity, cognitive function, and cardiometabolic risk. The investigators hypothesize that long-term intake of this diet will significantly potentiate the effects of a healthy lifestyle (physical activity and Mediterranean diet), constituting a powerful strategy to halt or even reverse the progression of several age-related processes related to adiposity, cardiometabolic health and cognition. The investigators further hypothesize that lifestyle intervention might modify the gut microbiota profile and that autologous fecal microbiota supplement derived from the time of maximal weight loss might halt the expected subsequent regain phase. The investigators will follow the participants with magnetic resonance imaging (MRI) that will include abdominal and hepatic fat, cardiac and anatomic/functional brain assessments. The investigators will perform cognitive tests and will measure changes in gut microbiota and sub-metabolomic profiling. The trial will be performed in an isolated workplace (the Nuclear Research Center) which holds an exclusive cafeteria that provides free, dietary -monitored, lunch, and an internal medical department. The exclusive nutritional profile of walnuts, with its relative high polyphenols content and unique composition, may benefit several health outcomes. Epidemiologic studies and RCTs suggest that walnuts consumption is associated with better weight status, adiposity measures and cardiometabolic state. However, some individuals avoid walnuts because they are calorie-dense, and fear that they will promote weight gain. Walnuts contain numerous well-characterized beneficial nutritional components, such as unsaturated fats, especially omega-3 fatty acids, dietary fibers, and high levels of vitamins and minerals. Among other well-recognized components, nuts are highly rich in polyphenols, mainly flavonoids. Polyphenols may potentially interact with physical activity and promote neurogenesis; a process that may significantly contribute to the brain's ageing process. Similarly, the polyphenol epigallocatechin-3-gallate (EGCG, a type of catechin found in green tea), was proposed to exert neuroprotective effects. New specific developed strain of duckweed [Wolffia globose, "Mankai"] , an aquatic plant, which might serve as a protein source and contains all the 9 essential and the 6 conditional amino acids. "Mankai" [(Generally recognized as safe (GRAS)] is a cultivated strain of Wolffia globosa, which is an aquatic plant, part of the family of plants known commonly as duckweeds. Duckweeds are very simple flowering aquatic plants, which float on or just beneath the surface of still or slow-moving bodies of water. There is a long history of the use of Wolffia species, in particular Wolffia Globosa, as food, especially in Southeast Asia: Burma, Laos and northern Thailand, where it has been used as a vegetable for many generations. The nutritional composition of "Mankai" has been determined and found to be high in protein, containing all the essential and conditionally essential amino acids, dietary fibers and several vitamins and minerals.

ELIGIBILITY:
Inclusion Criteria:

age >30 years with abdominal adiposity (waist circumference: men > 102 cm, women > 88 cm) or dyslipidemia (TG>150mg/dl and HDL-c <40mg/dL for men and <50mg/dL for women)

Exclusion Criteria:

Individuals who may not be able to partake in PA in the gym; TGs>400 mg/dL; serum creatinine>2 mg/dL; disturbed liver function; major illness that might require hospitalization; pregnant or lactating women; presence of active cancer, is receiving or received chemotherapy in the last three years; participation in another trial; participants who are treated with Coumadin (warfarin) - given its interaction with vitamin K and high level of this vitamin in "Mankai" green shake; pacemaker or platinum implant, because of the impossibility of MRI screening.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Abdominal fat | 18 months
  Changes in visceral fat (MRI)
Hepatic fat | 18 months
  Changes in hepatic fat (MRI)
Obesity | 6, 14, 18 months
  Changes in body weight and waist circumference

SECONDARY OUTCOMES:
Brain anatomy | 18 months
  Changes in hippocampus volume, diffusion Tensor Imaging (MRI)
Cognitive function-MRI | 18 months
  Changes in resting state connectivity (MRI, sub-study)
Cognitive function | 18 months
  cognitive tests
Cardiac state | 18 months
  Changes in cardiac anatomy (MRI, substudy)
Cardiac state | 18 months
  Changes in cardiac function (MRI, substudy)
Endothelial dysfunction | 18 months
  Changes endothelial function (ECG)
Lipid profile | 6 , 14 and 18 months
  Changes in lipid biomarkers (blood draw)
Glycemic control | 6 , 14 and 18 months
  Changes in glycemic biomarkers (blood draw)
Inflammatory state | 6 , 14 and 18 months
  Changes in inflammatory biomarkers (blood draw)
Metabolomic | 18 months
  Changes in sub-lipids (blood draw)
Metabolomic | 18 months
  Changes in sub-proteins ( blood draw)
Liver function (blood biomarkers) | 6 and 18 months
  Changes in liver function biomarkers (blood draw)
Genetic signature | baseline
  SNPs associated with fat distribution and visceral fat
Epigenetics | 18 months
  changes in mRNAs
Epigenetics | 18 months
  changes in genes' methylation
Well being | 18 months
  assessed by questionnaire
Fecal microbiota profile | 6, 14, 18 months
  Diversity Index as a key measure
24h- continuous glucose levels | 2 weeks
  24h dynamics of glucose using continuous glucose monitor. substudy

CONTACTS AND LOCATIONS:
Overall Officials: Iris Shai, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Nuclear research center Negev, Dimona, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein H, Pachter D, Goldberg Toren DT, Kamer O, Alufer L, Ebstein Karamani N, Chassidim Y, Shelef I, Rudich A, Yoel U, Ben-Arie G, Zelicha H, Yaskolka Meir A, Tsaban G, Bartal C, Bluher M, Stumvoll M, Ceglarek U, Isermann B, Qi L, Stampfer MJ, Hu FB, Shai I. How effective is rejoining a long-term weight loss program? The 5- and 10-year MRI-assessed Follow Interventions Trial (FIT) project. BMC Med. 2026 Jan 30. doi: 10.1186/s12916-026-04663-9. Online ahead of print. PMID 41612310
- [Derived] Pachter D, Yaskolka Meir A, Kaplan A, Tsaban G, Zelicha H, Rinott E, Levakov G, Finkelstein O, Shelef I, Salti M, Beyer F, Witte V, Kloting N, Isermann B, Ceglarek U, Riklin Raviv T, Bluher M, Stumvoll M, Wang DD, Hu FB, Stampfer MJ, Avidan G, Shai I. Serum Galectin-9 and Decorin in relation to brain aging and the green-Mediterranean diet: A secondary analysis of the DIRECT PLUS randomized trial. Clin Nutr. 2025 Oct;53:99-108. doi: 10.1016/j.clnu.2025.08.021. Epub 2025 Aug 23. PMID 40897150
- [Derived] Yaskolka Meir A, Tsaban G, Rinott E, Zelicha H, Schwarzfuchs D, Gepner Y, Rudich A, Shelef I, Bluher M, Stumvoll M, Ceglarek U, Isermann B, Kloting N, Keller M, Kovacs P, Qi L, Wang DD, Liang L, Hu FB, Stampfer MJ, Shai I. Individual response to lifestyle interventions: a pooled analysis of three long-term weight loss trials. Eur J Prev Cardiol. 2025 Nov 11;32(16):1660-1670. doi: 10.1093/eurjpc/zwaf308. PMID 40472282
- [Derived] Klein H, Zelicha H, Yaskolka Meir A, Rinott E, Tsaban G, Kaplan A, Chassidim Y, Gepner Y, Bluher M, Ceglarek U, Isermann B, Stumvoll M, Shelef I, Qi L, Li J, Hu FB, Stampfer MJ, Shai I. Visceral adipose tissue area and proportion provide distinct reflections of cardiometabolic outcomes in weight loss; pooled analysis of MRI-assessed CENTRAL and DIRECT PLUS dietary randomized controlled trials. BMC Med. 2025 Feb 4;23(1):57. doi: 10.1186/s12916-025-03891-9. PMID 39901232
- [Derived] Pachter D, Kaplan A, Tsaban G, Zelicha H, Meir AY, Rinott E, Levakov G, Salti M, Yovell Y, Huhn S, Beyer F, Witte V, Kovacs P, von Bergen M, Ceglarek U, Bluher M, Stumvoll M, Hu FB, Stampfer MJ, Friedman A, Shelef I, Avidan G, Shai I. Glycemic control contributes to the neuroprotective effects of Mediterranean and green-Mediterranean diets on brain age: the DIRECT PLUS brain-magnetic resonance imaging randomized controlled trial. Am J Clin Nutr. 2024 Nov;120(5):1029-1036. doi: 10.1016/j.ajcnut.2024.09.013. Epub 2024 Sep 14. PMID 39284453
- [Derived] Alufer L, Tsaban G, Rinott E, Kaplan A, Meir AY, Zelicha H, Ceglarek U, Isermann B, Bluher M, Stumvoll M, Stampfer MJ, Shai I. Long-term green-Mediterranean diet may favor fasting morning cortisol stress hormone; the DIRECT-PLUS clinical trial. Front Endocrinol (Lausanne). 2023 Nov 14;14:1243910. doi: 10.3389/fendo.2023.1243910. eCollection 2023. PMID 38034010
- [Derived] Kamer O, Rinott E, Tsaban G, Kaplan A, Yaskolka Meir A, Zelicha H, Knights D, Tuohy K, Fava F, Uwe Scholz M, Ziv O, Rubin E, Bluher M, Stumvoll M, Ceglarek U, Clement K, Koren O, Hu FB, Stampfer MJ, Wang DD, Youngster I, Shai I. Successful weight regain attenuation by autologous fecal microbiota transplantation is associated with non-core gut microbiota changes during weight loss; randomized controlled trial. Gut Microbes. 2023 Dec;15(2):2264457. doi: 10.1080/19490976.2023.2264457. Epub 2023 Oct 5. PMID 37796016
- [Derived] Yaskolka Meir A, Keller M, Hoffmann A, Rinott E, Tsaban G, Kaplan A, Zelicha H, Hagemann T, Ceglarek U, Isermann B, Shelef I, Bluher M, Stumvoll M, Li J, Haange SB, Engelmann B, Rolle-Kampczyk U, von Bergen M, Hu FB, Stampfer MJ, Kovacs P, Liang L, Shai I. The effect of polyphenols on DNA methylation-assessed biological age attenuation: the DIRECT PLUS randomized controlled trial. BMC Med. 2023 Sep 25;21(1):364. doi: 10.1186/s12916-023-03067-3. PMID 37743489
- [Derived] Zelicha H, Kloting N, Kaplan A, Yaskolka Meir A, Rinott E, Tsaban G, Chassidim Y, Bluher M, Ceglarek U, Isermann B, Stumvoll M, Quayson RN, von Bergen M, Engelmann B, Rolle-Kampczyk UE, Haange SB, Tuohy KM, Diotallevi C, Shelef I, Hu FB, Stampfer MJ, Shai I. The effect of high-polyphenol Mediterranean diet on visceral adiposity: the DIRECT PLUS randomized controlled trial. BMC Med. 2022 Sep 30;20(1):327. doi: 10.1186/s12916-022-02525-8. PMID 36175997
- [Derived] Rinott E, Meir AY, Tsaban G, Zelicha H, Kaplan A, Knights D, Tuohy K, Scholz MU, Koren O, Stampfer MJ, Wang DD, Shai I, Youngster I. The effects of the Green-Mediterranean diet on cardiometabolic health are linked to gut microbiome modifications: a randomized controlled trial. Genome Med. 2022 Mar 10;14(1):29. doi: 10.1186/s13073-022-01015-z. PMID 35264213
- [Derived] Kaplan A, Zelicha H, Yaskolka Meir A, Rinott E, Tsaban G, Levakov G, Prager O, Salti M, Yovell Y, Ofer J, Huhn S, Beyer F, Witte V, Villringer A, Meiran N, B Emesh T, Kovacs P, von Bergen M, Ceglarek U, Bluher M, Stumvoll M, Hu FB, Stampfer MJ, Friedman A, Shelef I, Avidan G, Shai I. The effect of a high-polyphenol Mediterranean diet (Green-MED) combined with physical activity on age-related brain atrophy: the Dietary Intervention Randomized Controlled Trial Polyphenols Unprocessed Study (DIRECT PLUS). Am J Clin Nutr. 2022 May 1;115(5):1270-1281. doi: 10.1093/ajcn/nqac001. PMID 35021194
- [Derived] Tsaban G, Yaskolka Meir A, Zelicha H, Rinott E, Kaplan A, Shalev A, Katz A, Brikner D, Bluher M, Ceglarek U, Stumvoll M, Stampfer MJ, Shai I. Diet-induced Fasting Ghrelin Elevation Reflects the Recovery of Insulin Sensitivity and Visceral Adiposity Regression. J Clin Endocrinol Metab. 2022 Jan 18;107(2):336-345. doi: 10.1210/clinem/dgab681. PMID 34643713
- [Derived] Yaskolka Meir A, Rinott E, Tsaban G, Zelicha H, Kaplan A, Rosen P, Shelef I, Youngster I, Shalev A, Bluher M, Ceglarek U, Stumvoll M, Tuohy K, Diotallevi C, Vrhovsek U, Hu F, Stampfer M, Shai I. Effect of green-Mediterranean diet on intrahepatic fat: the DIRECT PLUS randomised controlled trial. Gut. 2021 Nov;70(11):2085-2095. doi: 10.1136/gutjnl-2020-323106. Epub 2021 Jan 18. PMID 33461965
- [Derived] Tsaban G, Yaskolka Meir A, Rinott E, Zelicha H, Kaplan A, Shalev A, Katz A, Rudich A, Tirosh A, Shelef I, Youngster I, Lebovitz S, Israeli N, Shabat M, Brikner D, Pupkin E, Stumvoll M, Thiery J, Ceglarek U, Heiker JT, Korner A, Landgraf K, von Bergen M, Bluher M, Stampfer MJ, Shai I. The effect of green Mediterranean diet on cardiometabolic risk; a randomised controlled trial. Heart. 2021 Jun 11;107(13):1054-1061. doi: 10.1136/heartjnl-2020-317802. PMID 33234670
- [Derived] Rinott E, Youngster I, Yaskolka Meir A, Tsaban G, Zelicha H, Kaplan A, Knights D, Tuohy K, Fava F, Scholz MU, Ziv O, Rubin E, Tirosh A, Rudich A, Bluher M, Stumvoll M, Ceglarek U, Clement K, Koren O, Wang DD, Hu FB, Stampfer MJ, Shai I. Effects of Diet-Modulated Autologous Fecal Microbiota Transplantation on Weight Regain. Gastroenterology. 2021 Jan;160(1):158-173.e10. doi: 10.1053/j.gastro.2020.08.041. Epub 2020 Aug 26. PMID 32860791
- [Derived] Yaskolka Meir A, Tsaban G, Zelicha H, Rinott E, Kaplan A, Youngster I, Rudich A, Shelef I, Tirosh A, Brikner D, Pupkin E, Sarusi B, Bluher M, Stumvoll M, Thiery J, Ceglarek U, Stampfer MJ, Shai I. A Green-Mediterranean Diet, Supplemented with Mankai Duckweed, Preserves Iron-Homeostasis in Humans and Is Efficient in Reversal of Anemia in Rats. J Nutr. 2019 Jun 1;149(6):1004-1011. doi: 10.1093/jn/nxy321. PMID 30915471